CLINICAL TRIAL: NCT06459570
Title: Efficacy of VR Based Sword Fighting Exercises to Improve Upper Body Movements in Hemiplegic Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/729
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hemiplegic Gait
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality based exercises (Experimental)
  Interventions: Behavioral: Virtual reality based exercises
- standard physical therapy (Other)
  Interventions: Other: standard physical therapy

INTERVENTIONS:
Behavioral: Virtual reality based exercises — one experimental group with Virtual reality-based exercises. Subjects in the VR-based exercises will receive 12 sessions of the VR-based exercises treatment, administered four times a week over 3 weeks, with each session lasting approximately 60 minutes.
  Arms: Virtual reality based exercises
Other: standard physical therapy — "Second control group with standard physical therapy and occupational therapy treatment.Subjects in the control group will receive 12 sessions of physical therapy treatment involving passive and active range of motion exercises, muscle strengthening, and therapeutic stretching, administered four times a week over a span of 3 weeks, with each session lasting approximately 60 minutes.
  Arms: standard physical therapy

SUMMARY:
this thesis endeavors to shed light on the efficacy of VR-based sword-fighting exercises as a rehabilitation tool for improving upper body movement in hemiplegic patients.

DETAILED DESCRIPTION:
By amalgamating clinical insights, technological advancements, and theoretical frameworks, this research aims to contribute to the growing body of knowledge in neurorehabilitation and pave the way for innovative, effective, and engaging interventions to enhance the lives of individuals affected by hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years
* First clinical stroke, ischemic or hemorrhagic, with diagnosis of stroke confirmed on CT/MRI brain scan.
* Less than 6 weeks after stroke onset
* Upper limb weakness of Medical Research Council (MRC) motor power of grade 2-4 motor power in either the shoulder, elbow or the fingers of the hemiplegic upper extremity
* Subject can understand simple instructions and learn

Exclusion Criteria:

* Recurrent stroke
* History of epilepsy
* Presence of arthritis or pain in the affected upper limb restricting repetitive exercises
* Severe aphasia or cognitive impairment, or other psychiatric illnesses that limit the ability to participate or give consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment of upper limb (FMA) | 12 Months
  This measures upper limb impairment and scores from 0 to 66, the higher the score, the less the impairment. The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation, and joint functioning in patients with post-stroke hemiplegia.
Action Research Arm Test (ARAT) | 12 months
  This measures arm and hand function and ranges from 0 to 57, the higher the score, the better the upper limb function. The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No